CLINICAL TRIAL: NCT02245789
Title: Does the Use of a Videolaryngoscope Modifies Anesthetic Induction ?
Acronym: MGM-PicRemi
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2013/43; 2013-A01308-37 (Other: ANSM)
Record Dates: First submitted 2014-09-04; First posted 2014-09-22 (Estimated); Last update posted 2016-10-31 (Estimated); Status verified 2016-10

CONDITIONS: Tracheal Intubation
MeSH Terms: interventions — Intubation, Intratracheal; Propofol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Macintosh laryngoscope (Active Comparator): Tracheal intubation will be performed using a Macintosh laryngoscope. All patients will received propofol and remifentanil anesthesia.
  Interventions: Procedure: Tracheal intubation; Drug: Propofol and remifentanil anesthesia
- McGrath Mac videolaryngoscope (Experimental): Tracheal intubation will be performed using a McGrath Mac videolaryngoscope. All patients will received propofol and remifentanil anesthesia.
  Interventions: Procedure: Tracheal intubation; Drug: Propofol and remifentanil anesthesia

INTERVENTIONS:
Procedure: Tracheal intubation — Tracheal intubation will be performed using a Macintosh laryngoscope or a McGrath Mac videolaryngoscope
Drug: Propofol and remifentanil anesthesia — The standardized anesthetic procedure used a closed-loop anesthesia system with bispectral index as control variable and with two proportional-differential control algorithms, one for propofol target-controlled infusion system and one for remifentanil target-controlled infusion system.

SUMMARY:
Videolaryngoscopes become widely used. The aim of this study is to compare anesthetic induction when patients are tracheally intubated using a MacGraph Mac videolaryngoscope or a conventional MacIntosh laryngoscope.

Tracheal intubation induces a nociceptive stimulation. Hypothesis is that the use of a videolaryngoscope induces a less pronounced nociceptive stimulation and, consequently, that it modifies the anesthetic drugs requirement. .

DETAILED DESCRIPTION:
All patients will received a standardized anesthetic procedure : combined closed-loop anesthesia system using bispectral index as control variable and two proportional-differential control algorithms, a propofol and a remifentanil target-controlled infusion system. The effectiveness of such a closed-loop anesthesia system has been demonstrated in a prospective, randomized study.

Patients will be randomized in two groups : intubation using a conventional MacIntosh laryngoscope or intubation using a videolaryngoscope.

If our hypothesis is confirmed, the required concentration of remifentanil, an opioid agent, will be reduced in the group using a videolaryngoscope.

ELIGIBILITY:
Inclusion Criteria:

* patient scheduled for a general anesthesia with orotracheal intubation

Exclusion Criteria:

* predictable risk of difficult mask ventilation or of difficult tracheal intubation
* necessity of a rapid sequence induction
* contra-indication to the use of the automated administration of propofol and of remifentanil
* contra-indication to the use of atracurium
* Otolaryngology, thoracic surgery, or intracranial surgery

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-09; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Required dose of opioid to counteract nociceptive stimulation | 1 hour
  Tracheal intubation induces a nociceptive stimulation. Hypothesis is that the use of a videolaryngoscope induces a less pronounced nociceptive stimulation and, consequently, that the required maximal concentration of remifentanil is lower than when a standard laryngoscope is used.

SECONDARY OUTCOMES:
Characteristics of anesthesia | one hour
  Peak concentration of propofol
Characteristics of anesthesia | one hour
  doses of propofol and of remifentanil (from beginning of the induction to 5 minutes after tracheal intubation)
Characteristics of anesthesia | one hour
  values of bispectral index (from beginning of the induction to 5 minutes after tracheal intubation)
Characteristics of tracheal intubation | one hour
  time to obtain the first capnogram
Characteristics of tracheal intubation | one hour
  visualization of the glottis (score of Cormak and Lehane modified by Yentis, POGO score
Characteristics of tracheal intubation | one hour
  use of alternative techniques for intubation
Characteristics of tracheal intubation | one hour
  esophageal intubation
Characteristics of tracheal intubation | one hour
  incidence of arterial oxygen desaturation (SpO2 <92%)
Characteristics of tracheal intubation | one hour
  hemodynamic effects of induction and tracheal intubation
Complications of intubation | one day
  Throat pain and hoarseness
Ergonomic evaluation of the device | one hour
  questionnaire Qusi

CONTACTS AND LOCATIONS:
Overall Officials: Michel Chandon, MD, Principal Investigator — Hopital Foch
Locations (2):
- France (2):
  - Institut Hospitalier Franco-Britannique, Levallois-Perret, Hauts de Seine
  - Hopital Foch, Suresnes, Hauts de Seine

REFERENCES:
- [Background] Liu N, Chazot T, Hamada S, Landais A, Boichut N, Dussaussoy C, Trillat B, Beydon L, Samain E, Sessler DI, Fischler M. Closed-loop coadministration of propofol and remifentanil guided by bispectral index: a randomized multicenter study. Anesth Analg. 2011 Mar;112(3):546-57. doi: 10.1213/ANE.0b013e318205680b. Epub 2011 Jan 13. PMID 21233500
- [Derived] Ing R, Liu N, Chazot T, Fessler J, Dreyfus JF, Fischler M, Le Guen M. Nociceptive stimulation during Macintosh direct laryngoscopy compared with McGrath Mac videolaryngoscopy: A randomized trial using indirect evaluation using an automated administration of propofol and remifentanil. Medicine (Baltimore). 2017 Sep;96(38):e8087. doi: 10.1097/MD.0000000000008087. PMID 28930848